CLINICAL TRIAL: NCT05309382
Title: Development of Non-invasive Cell-free DNA to Supplant Invasive Biopsy in Heart Transplant
Brief Title: Development of Non-invasive Cell-free DNA to Supplant Invasive Biopsy in Heart Transplantation
Acronym: DEFINE-HT
Status: Completed | Type: Observational
Sponsor: Natera, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 22-062-TRP
Record Dates: First submitted 2022-03-25; First posted 2022-04-04 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Heart Transplant
Keywords: Prospera; dd-cfDNA; Heart; Transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Prospera — Monthly testing and results provided

SUMMARY:
This is a prospective, multicenter observational, unblinded, longitudinal cohort study. Subjects will be enrolled into the study prior to or at the time of heart transplantation. All subjects will follow the center's standard of care surveillance schedule. Blood samples will be collected for Prospera testing at the time any surveillance or for-cause testing, which may include endomyocardial biopsy (EMB), echocardiography or other cardiac imaging studies, and/or molecular testing, is performed.

DETAILED DESCRIPTION:
Subjects will undergo surveillance monitoring for rejection per the institution's standard clinical care schedule after transplant. Surveillance procedures may include EMB, imaging such as echocardiography, and/or molecular testing. Surveillance is expected to occur at this approximate schedule during the 12 months post-transplant:

* Weekly during month 1
* Every other week months 2-3
* Monthly during months 4-6
* Every 1-3 months during months 7-12

For-cause testing for rejection will be performed as clinically indicated and per the institution's standard clinical care. Prospera testing will be performed at the time each standard of care (SOC) rejection surveillance procedure and at the time of each for-cause testing for rejection. Prospera test results will be provided to the clinical team.

Additional blood samples for research only will be collected at the time of each Prospera blood sample collection. Results of testing performed on research blood samples will not be returned to investigators for use in clinical care.

Study central laboratory or central review for research purposes will include:

1. Central pathology review (all EMBs, includes for-cause EMBs).
2. Central echocardiography review at day 30 (± 14 days), month 6 (± 30 days) and month 12 (± 30 days) post-transplant.
3. Central testing of PRA/DSA pre-transplant (between enrollment and transplant), at day 30 (± 14 days), month 6 (± 30 days) and month 12 (± 30 days) post-transplant.

Central pathology and echocardiography review will be performed using uploaded images obtained from procedures performed as part of routine clinical care. Central pathology review, central echocardiography review and central laboratory PRA/DSA are for research purposes; these data will be reviewed during the analysis phase of the study and results will not be returned to investigators for use in clinical care.

The study period will start at enrollment and conclude with the final visit at 12 months +/- 30 days post-transplant.

This study will generate additional preliminary data to be used in the design and implementation of a subsequent confirmatory clinical utility trial.

The primary objectives are to:

1. Describe the association between Prospera dd-cfDNA measures and other diagnostic tests used to detect heart allograft rejection and/or injury, including histology, echocardiography and DSA, in the first post-transplant year
2. Inform rates of clinical outcomes in a contemporary cohort of adult heart transplant recipients to determine power for a future randomized, controlled clinical trial.

The secondary objectives are to determine:

1. The performance characteristics of the Prospera dd-cfDNA assay to discriminate biopsyproven acute rejection (AR).
2. The performance characteristics of the Prospera dd-cfDNA assay to discriminate acute cellular rejection (ACR).
3. The performance characteristics of the Prospera dd-cfDNA assay to discriminate antibody mediated rejection (AMR).
4. The association between dd-cfDNA levels and donor specific antibodies.
5. The association between dd-cfDNA levels and allograft dysfunction as measured by echocardiography.
6. The association between dd-cfDNA levels and allograft hemodynamics as measured by right heart catheterization.
7. The association between dd-cfDNA levels and future adverse clinical outcomes.
8. The effect of treatment for rejection on dd-cfDNA.
9. The variability of dd-cfDNA by patient characteristics, including race and gender.
10. The variability of dd-cfDNA across donor-recipient characteristics, including gender and race mismatch.
11. The association between dd-cfDNA (fraction and absolute level) and predicted heart mass.
12. The association between dd-cfDNA levels and time since transplant.
13. The association between dd-cfDNA levels and rejection with hemodynamic compromise (requiring inotropes and/or mechanical circulatory support).
14. The association between dd-cfDNA levels and incidence of cardiac allograft vasculopathy at one year.
15. The association between dd-cfDNA levels and different regimens of immunosuppression

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older at the time of signing informed consent.
2. Undergoing transplant evaluation or currently on the heart transplant waiting list and expected to receive a heart transplant.
3. Able to read, understand, and provide written informed consent.
4. Able and willing to comply with the study visit schedule, study procedures, and study requirements.

Exclusion Criteria:

1. Concurrent multiple solid organ or tissue transplants.
2. Prior history of any organ or cellular transplantation.
3. Pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart transplant rejection
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
Primary Molecular Endpoint | 1 year
  Percent and quantity of donor-derived cell-free DNA (dd-cfDNA) measured via the Prospera test.
Primary clinical endpoint* | 12 months
  Incidence of the composite endpoint of treated rejection, graft dysfunction, re-transplantation, or death at 12 months after transplant.
  *Clinical endpoints are defined as follows:
  1. Treated rejection: treated biopsy proven rejection (ISHLT ACR Grade ≥ 2R or AMR Grade ≥ pAMR1) or biopsy-negative rejection treated with pulse-dose steroids, monoclonal antibodies, plasmapheresis and/or intravenous immunoglobulin (IVIg).
  2. Graft dysfunction: left ventricular ejection fraction (LVEF) decline >10% from baseline and < 50% absolute LVEF by echocardiography.
  3. Re-transplantation: being listed for re-transplant or being re-transplanted.
  4. Death due to any cause.

SECONDARY OUTCOMES:
Secondary Endpoints | 12 months
  The secondary endpoints are:
  1. Incidence of the individual components of the primary composite endpoint at 12 months after transplant.
  2. The incidence at 12 months of:
     1. Rejection with hemodynamic compromise (requiring inotropes and/or mechanical circulatory support);
     2. The development of de novo donor specific antibodies;
     3. Cardiac allograft vasculopathy.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Olymbios, MD, Study Director — Natera, Inc.; Palak Shah, MD, Principal Investigator — Inova Health Care Services; Josef Stehlik, MD, Study Chair — University of Utah
Locations (9):
- United States (9):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - Mayo Clinic, Jacksonville, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Utah, Salt Lake City, Utah
  - Inova Heart and Vascular Institute, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: No